CLINICAL TRIAL: NCT06058780
Title: Safety and Efficacy of Implantable Collamer Lens Versus Implantable Phakic Lens IPCL in Myopic Patients; A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Akram Fekry Elgazzar, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICL vs IPCL
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Lenses, Intraocular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implantable Collamer Lens (ICL) (Active Comparator)
  Interventions: Procedure: Implantable Collamer Lens (ICL)
- Implantable Intraocular Lens (IPCL) (Active Comparator)
  Interventions: Procedure: Implantable Intraocular Lens (IPCL)

INTERVENTIONS:
Procedure: Implantable Collamer Lens (ICL) — Phakic intraocular lenses (pIOL) have proven to be a great alternative to corneal refractive surgery in certain situations. They offer several advantages over corneal techniques, such as being suitable for high myopes and causing relatively fewer higher-order aberrations
  Arms: Implantable Collamer Lens (ICL)
Procedure: Implantable Intraocular Lens (IPCL) — The IPCL offers a distinct economic advantage as the cost of the IPCL implant is only 2. times that of the ICL implant. Moreover, the IPCL can correct higher degrees of myopia, up to -30. D, compared to the maximum correction of -18. D provided by the ICL.
  Arms: Implantable Intraocular Lens (IPCL)

SUMMARY:
Phakic intraocular lenses (pIOL) have proven to be a great alternative to corneal refractive surgery in certain situations. They offer several advantages over corneal techniques, such as being suitable for high myopes and causing relatively fewer higher-order aberrations. In addition, pIOLs have been shown to provide better retinal image magnification and higher contrast sensitivity compared to laser in situ keratomileusis, regardless of whether the myopia is low or high.

ELIGIBILITY:
Inclusion Criteria:

* myopia of more than 6 diopter

Exclusion Criteria:

* unstable refraction
* unstable refraction

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
UCVA | Baseline
  Uncorrected Visual Acuity measured in decimal
UCVA | 3 months postoperative
  Uncorrected Visual Acuity measured in decimal
UCVA | 6 months postoperative
  Uncorrected Visual Acuity measured in decimal
UCVA | 12 months postoperative
  Uncorrected Visual Acuity measured in decimal
BCVA | Baseline
  Best corrected Visual Acuity measured in decimal
BCVA | 3 months postoperative
  Best corrected Visual Acuity measured in decimal
BCVA | 6 months postoperative
  Best corrected Visual Acuity measured in decimal
BCVA | 12 months postoperative
  Best corrected Visual Acuity measured in decimal
Refraction | Baseline
  Preoperative refractive error measured in spherical equivalent
Refraction | 3 months postoperative
  postoperative refractive error measured in spherical equivalent
Refraction | 6 months postoperative
  postoperative refractive error measured in spherical equivalent
Refraction | 12 months postoperative
  postoperative refractive error measured in spherical equivalent

CONTACTS AND LOCATIONS:
Locations (1):
- Akram Fekry Elgazzar, Damietta, Egypt